CLINICAL TRIAL: NCT03203044
Title: Impact of Soylent Consumption on Human Microbiome Composition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Responsible Party: Principal Investigator, Adam P. Arkin, Professor, University of California, Berkeley
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: soylentmicrobiomeproject
Record Dates: First submitted 2017-06-27; First posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Gut Microbiota
Keywords: Dietary Intervention

STUDY DESIGN:
Intervention Model Description: Participants are separated into two diet arms. The regular diet arm remains on a self-reported regular diet for the duration of the study. The Soylent diet arm maintains a regular diet for two days, switches to an all Soylent and water diet for four days, and returns to a regular diet for four days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular Diet Arm (No Intervention): Maintains a regular diet for the duration of the study.
- Soylent Diet Arm (Experimental): Receives a Soylent dietary intervention on days 3-6 of the study.
  Interventions: Other: Soylent and water diet

INTERVENTIONS:
Other: Soylent and water diet — A diet of five servings of Soylent 2.0 liquid meal-replacement drink per day and water as needed.
  Arms: Soylent Diet Arm

SUMMARY:
Soylent 2.0 is a popular meal replacement drink that is used to supplement or replace one's regular diet. Soylent is designed to fully fulfill one's nutritional needs, but its impact on the human microbiome remains unknown. This study aims to track the composition of participants' gut microbiomes before, during, and after Soylent consumption to more holistically understand its impact on microbiome health. We predict that a short term Soylent-based diet will induce observable and reversible changes to participants' gut microbiomes.

DETAILED DESCRIPTION:
After collecting this preliminary information, main study participants will be chosen based on our described inclusion/exclusion criteria. We will distribute eight fecal sampling kits to each participant in preparation for the study. The study duration is 10 days and consists of three phases:

In Phase A, participants will adhere to their regular diet for two days. This initial condition provides a baseline of each participant's unique microbiome, acting as an internal control.

In Phase B, a subset of the participants, which will be chosen by random drawing from a box, will switch to an all-Soylent diet. During this phase, they will consume five bottles of Soylent 2.0 daily for four days (one for breakfast, two for lunch, and two for dinner), fully meeting a 2000kcal diet and all recommended nutritional daily values. The remaining participants will retain their regular diets for four days. These individuals act as a control for the daily variance of microbiome fluctuations.

In Phase C, participants will return to their regular diets for four days, after which the study will conclude.

For the duration of the study, participants will log their diets and bowel movements electronically on a daily basis. A printout of the Bristol Stool Chart will be provided at the beginning of the study to each participant. Each entry will be logged through a Google Form and labeled with each individual's participant ID, which will link them to their responses. The link will include name, email, and phone number. The completed forms are only accessible through a single Google account, which is password protected, encrypted, and only accessible by the investigators. In addition, participants will sample their microbiomes using the uBiome gut kits on the following days: 1, 2, 3, 4, 5, 6, 7, and 10. Sampling is done by swabbing used toilet paper after bowel movements. Participants will seal the samples in the kits and mail them to uBiome with the included prepaid postage. The investigators will not come into direct contact with any of the samples.

All electronic logs and samples will be labeled with each participant's unique participant ID. The link between each participant and their sample kits will be maintained on the participant reference sheet kept by the researchers. uBiome will not have access to this link.

Once all data in the study has been received, the participant reference sheet will be shredded and all of the data will become unidentifiable. While Soylent has no documented instances of causing physical complications to consumers, if any participant feels unwell during any point in the study, they are encouraged to cease participation and contact their primary care doctor for guidance.

Results from the uBiome gut kits will be received in about four to six weeks. uBiome will share the data individually with each participant (if participants chose to create an account and register their kits as stated above) and in bulk with the researchers. For participants that did not register their kits with uBiome, the data generated from those participants will only be sent to the researchers. The data consists of sequencing data labeled with each kit's serial number. We will then correlate our electronic log data with the uBiome sample data for further analysis. The data generated in this study is in no way intended for medical diagnosis of any kind. uBiome's website states the following: "It's important to be aware that uBiome is designed to be a tool for personal research, NOT a diagnostic tool. You won't find any predictions about your future health. And your results will not diagnose any medical condition."

ELIGIBILITY:
Inclusion Criteria:

* The subject population will consist of undergraduate UC Berkeley students.

Exclusion Criteria:

* Dietary allergies or sensitivities to Soylent 2.0 ingredients
* Vulnerable individuals as defined by Committee for Protection of Human Subjects guidelines
* Individuals with health issues
* Individuals who take antibiotics, probiotics, alcohol, or supplements.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2016-11-16 (Actual); Study Completion 2016-11-16 (Actual)

PRIMARY OUTCOMES:
Changes to gut microbiome composition as a result of an interventional Soylent diet | Days 3-6 of the study

CONTACTS AND LOCATIONS:
Overall Officials: Adam P Arkin, PhD, Principal Investigator — Professor

IPD SHARING:
Plan to Share IPD: Yes
Bacterial DNA sequencing data from collected fecal samples will be shared in a public repository. Sample labels will be deidentified.